CLINICAL TRIAL: NCT06945406
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY4057996 in Healthy Participants and Participants With Type 1 and Type 2 Diabetes
Brief Title: A Study of LY4057996 in Healthy Participants and Participants With Type 1 and Type 2 Diabetes
Acronym: YKAA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 27329; 2024-519151-28-00 (EU CTIS Number); J6B-MC-YKAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parts A and C are sequential: Part B is crossover
Who Masked: Participant, Investigator
Masking Description: Part A is Double-Blinded, Parts B and C are Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- LY4057996 Part A (Cohorts A1-A5) (Experimental): LY4057996 administered subcutaneously (SC) and/or intravenously (IV)
  Interventions: Drug: LY4057996 SC; Drug: LY4057996 IV
- Placebo Part A (Cohort A1-A5) (Placebo Comparator): Placebo administered SC and/or IV
  Interventions: Drug: Placebo SC; Drug: Placebo IV
- LY4057996 Part B (Experimental): LY4057996 administered SC
  Interventions: Drug: LY4057996 SC
- LY4057996 Part C (Experimental): LY4057996 and interventions of pre-study basal insulin and Lispro administered SC
  Interventions: Drug: LY4057996 SC; Drug: Lispro SC; Drug: Pre-study basal insulin SC
- Degludec Part A (Cohort A2-A5) (Active Comparator): Degludec administered SC and/or IV
  Interventions: Drug: Degludec SC; Drug: Degludec IV
- Degludec Part B (Active Comparator): Degludec administered SC
  Interventions: Drug: Degludec SC

INTERVENTIONS:
Drug: LY4057996 SC — Administered SC
  Arms: LY4057996 Part A (Cohorts A1-A5); LY4057996 Part B; LY4057996 Part C
Drug: LY4057996 IV — Administered IV
  Arms: LY4057996 Part A (Cohorts A1-A5)
Drug: Placebo SC — Administered SC
  Arms: Placebo Part A (Cohort A1-A5)
Drug: Placebo IV — Administered IV
  Arms: Placebo Part A (Cohort A1-A5)
Drug: Degludec SC — Administered SC
  Arms: Degludec Part A (Cohort A2-A5); Degludec Part B
Drug: Lispro SC — Administered SC
  Arms: LY4057996 Part C
Drug: Degludec IV — Administered IV
  Arms: Degludec Part A (Cohort A2-A5)
Drug: Pre-study basal insulin SC — Administered SC
  Arms: LY4057996 Part C

SUMMARY:
The purpose of this study is to evaluate how well LY4057996 is tolerated and what side effects may occur in healthy participants and participants with Type 1 and Type 2 Diabetes. The study drug will be administered either subcutaneously (SC) (under the skin) or intravenously (IV) (into a vein in the arm). Blood tests will be performed to check how much LY4057996 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last 11 weeks for Part A1-A2, 4 weeks for A3-A5, 6 weeks for Part B and 7 weeks for Part C, all approximations, excluding a screening period.

ELIGIBILITY:
Inclusion Criteria:

Part A for Healthy Participants:

* Are overtly healthy as determined by medical evaluation, including medical history, physical exam, laboratory tests, and cardiac screening assessment

Part A for Type 2 Diabetes (T2DM) Participants:

* Are participants with T2DM diagnosed greater than 1 year before enrollment,
* On basal insulin therapy, insulin glargine, or insulin degludec, greater than 10 units per day for at least 6 months (for Cohort 5 only)
* Glycated hemoglobin (HbA1c) 6.5% to 9.5% inclusive at screening

Part B

* Have Type 1 Diabetes (T1D) for at least 1 year with a fasting C-peptide level of 0.20 nanomole per liter (nmol/L) or less or non-fasting C-peptide level of 0.30 nmol/L or less at screening
* HbA1c 6% to 8.5% inclusive at screening

Part C

* Have T1D for at least 1 year with a fasting C-peptide level of 0.20 nanomole per liter (nmol/L) or less or non-fasting C-peptide level of 0.30 nmol/L or less at screening
* HbA1c 6 to 8% inclusive at screening

All Parts

* Have blood pressure of less than 140/90 millimeters of mercury (mmHg) for healthy participants or 150/90 mmHg for participants with diabetes and pulse rate of less than 90 beats per minute (bpm) (supine)
* No hypoglycemia unawareness for all Type 1 and Type 2 Diabetes participants

Exclusion Criteria:

* Have had more than 1 emergency room visit or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis) within 6 months prior to screening
* Have had any episodes of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within the 6 months prior to screening

All Parts

* Cardiovascular: no significant history of cardiovascular disease (CVD)
* Gastrointestinal: have gastroparesis or have undergone gastric surgery
* Hepatic: have acute or chronic hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) and Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 47 Weeks)
  A summary of SAEs and AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY4057996 | Baseline to Study Completion (Up to 47 Weeks)
  PK: AUC of LY4057996
PK: Maximum Concentration (Cmax) of LY4057996 | Baseline to Study Completion (Up to 47 Weeks)
  PK: Cmax of LY4057996
Pharmacodynamic (PD): Change from Baseline in Fasting Glucose | Baseline to Study Completion (Up to 47 Weeks)
  PD: Change from Baseline in Fasting Glucose
PD: AUC of Glucose Infusion Rate (GIR) | Baseline Up to 10 weeks
  PD: AUC of GIR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4057996 in Healthy Participants and Participants With Type 1 and Type 2 Diabetes — https://trials.lilly.com/en-US/trial/599655